CLINICAL TRIAL: NCT04768374
Title: Effects of Virtual Reality on Cerebral Palsy; A Single-blind, Randomized Control Study: 3 Months Follow-up
Brief Title: Effects of Virtual Reality on Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Orkun Tahir Aran, PhD., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/ 2020- 214
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Enrolled into 12 week VR intervention with Microsoft Kinect (twice a week, for 45 minutes) and conventional occupational therapy.
  Interventions: Other: Virtual Reality with Kinect; Other: Conventional Occupational Therapy (COT)
- Control group (Active Comparator): Control group only received conventional occupational therapy for 12 weeks
  Interventions: Other: Conventional Occupational Therapy (COT)

INTERVENTIONS:
Other: Virtual Reality with Kinect — In the study it was conducted a 12 week-intensive VR intervention (twice a week, 45 minutes each) and compared the results in the 12th week to investigate the effects of rehabilitation and follow-up assessments were made in the 16th and 24th weeks. From the beginning of the VR intervention, each game was played in equal durations by each participant. However, the difficulty of the games varied depending on the child's performance.
  Microsoft Kinect Games-Carnival Games was used as VR intervention. In meeting held with the authors to determine which games would be used in the VR program, 5 games were chosen and the remaining games were removed from the program because of their similar contents.
  Arms: VR group
Other: Conventional Occupational Therapy (COT) — The COT based on neurodevelopmental treatment was carried out by the same occupational therapist. The treatment goals aimed at increasing the use of participant's extremities and improving the independence in ADL. The activities in the treatment were chosen in view of children's motor skills and daily living activities such as getting dressed, solving puzzles, and writing etc.
  Both groups received COT while the control group received COT only for 12 weeks.

SUMMARY:
Virtual reality (VR), is one of the most popular approaches to Cerebral Palsy (CP) rehabilitation and has been used in rehabilitation field for 30 years. VR is provided via a computer or a game console, and players interact with real-like objects . Using a VR interface as a rehabilitation tool increases the fun received by the client which, in turn, increases the participation of the client to the rehabilitation sessions.

This is a study that focused on long-term effects of Virtual reality (VR) intervention on motor skills and activities of daily living (ADL) independence of children with CP.

ELIGIBILITY:
Inclusion Criteria:

* had to be 7 to 12 years-old,
* to be diagnosed with CP,
* to get 1 or 2 from Gross Motor Functioning Classification System,
* to get a score of 1 to 3 from Manual Ability Classification System,
* to score at least 23 from Mini Mental State Examination - children edition,
* to be able to follow verbal instructions, and
* to have the

Exclusion Criteria:

* having any surgical operation and/or botulinum toxin injection in last 6 months,
* having any visual and hearing diseases that may affect using VR, and
* participating in any other rehabilitation programs (such as physiotherapy, speech therapy, psychotherapy etc.),
* having ataxic and/or dyskinetic symptoms.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Independence in Activities of Daily living (assessed with Abilhand-kids) | Baseline, 12th week (end of intervention), 24th and 36th week(follow up)
  ABILHAND-Kids is a scale that was developed to evaluate activities of daily living (ADL) requiring upper limb usage of children aged between 6-15 years
Change in motor proficiency( assessed with Bruninsk-Oseretsky Test of Motor Proficiency 2-Brief Form (BOT2-BF)) | Baseline, 12th week (end of intervention), 24th and 36th week(follow up)
  BOT2-BF is a test that evaluates motor proficiency and allows therapists to compare results with specified norm values

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No